CLINICAL TRIAL: NCT04859777
Title: A Phase 1/1b Study of MPT-0118 as Monotherapy and in Combination With Pembrolizumab in Subjects With Advanced or Metastatic Refractory Solid Tumors
Brief Title: A Study of MPT-0118 in Subjects With Advanced or Metastatic Refractory Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monopteros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MPT-0118-101
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Solid Tumor, Adult; Advanced Solid Tumor; Advanced Cancer; Metastatic Cancer; Refractory Cancer
Keywords: MALT1 inhibitor
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Part A: Each dose-escalation cohort will initially recruit single-subject cohorts until a subject has a Grade 2 or greater adverse event (AE) during the DLT period considered at least possibly related to MPT-0118, at which time 2 additional subjects will be enrolled in that cohort, and a 3 + 3 design will subsequently be utilized.
  Part B: Each dose-escalation cohort will initially recruit 3 patients to receive MPT-0118 + pembrolizumab in a standard 3+3 design; the cohort will be expanded in the event of a DLT.
  Part C: Once the RP2D has been established for MPT-0118 monotherapy and combination therapy with MPT-0118 + pembrolizumab, expansion cohorts will be enrolled to further evaluate combination therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: (Experimental): Dose-escalation oral MPT-0118 BID
  Interventions: Drug: MPT-0118
- Part B: (Experimental): Dose-escalation oral MPT-0118 BID + pembrolizumab (IV)
  Interventions: Drug: MPT-0118 + pembrolizumab
- Part C: (Experimental): Dose-expansion oral MPT-0118 BID + pembrolizumab (IV)
  Interventions: Drug: MPT-0118 + pembrolizumab

INTERVENTIONS:
Drug: MPT-0118 — MPT-0118 is an inhibitor of MALT1 protease
  Arms: Part A:
Drug: MPT-0118 + pembrolizumab — MPT-0118 is an inhibitor of MALT1 protease; pembrolizumab is a PD-1 inhibitor
  Arms: Part B:; Part C:

SUMMARY:
This is a Phase 1/1b open-label, dose-escalation, and cohort expansion study with BID (tablet) oral dose of MPT-0118 in subjects with advanced or metastatic refractory solid tumors.

The study will be conducted in 3 parts:

* Part A: MPT-0118 dose-escalation
* Part B: MPT-0118 dose-escalation in combination with pembrolizumab
* Part C: Cohort expansion of MPT-0118 in combination with pembrolizumab

DETAILED DESCRIPTION:
MPT-0118 will be administered orally twice daily (BID). Pembrolizumab will be administered intravenously (IV) at a dose of 200 mg every 3 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a histologically- or cytologically-diagnosed solid tumor which is advanced or metastatic and which has progressed on or following at least one systemic therapy regimen administered for advanced or metastatic disease or for which no approved therapy exists. Subject's prior treatment should include all approved regimens that have demonstrated a survival advantage for the subject's disease, stage, and line of therapy.
2. Is aged ≥18 years at the time of signing the ICF
3. Has provided written informed consent
4. Has an ECOG Performance Status of 0 or 1
5. Has measurable disease per RECIST 1.1
6. Has an adequate tumor sample.
7. Has adequate liver, renal, hematologic, pulmonary, cardiac, and coagulation function.
8. Has a negative serum pregnancy test (for women of child-bearing potential) at Screening and a negative urine pregnancy test on Day 1 prior to the first dose of MPT 0118
9. Ability to swallow and retain and absorb oral medications in tablet or crushed form orally or via feeding tube (e.g., nasogastric feeding tube or percutaneous endoscopic gastrostomy feeding tube)

Key Exclusion Criteria:

1. Has received cytotoxic chemotherapy, biologic agent, investigational agent, checkpoint inhibitors, or radiation therapy ≤3 weeks prior to the first dose of MPT-0118
2. Has received small-molecule kinase inhibitors or hormonal agents ≤14 days prior to the first dose of MPT-0118
3. Has been previously treated with a MALT1 inhibitor
4. Has clinically significant AEs that have not returned to baseline or ≤Grade 1 based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
5. Has received systemic immunosuppressive agents within 14 days of the first dose of MPT-0118
6. Has undergone major surgery ≤6 weeks or minor surgery ≤14 days prior to the first dose of MPT-0118
7. Has clinically significant intercurrent disease
8. Part B and Part C: Has previously been treated with PD-1, PD-L1, or CTLA-4 inhibitors and required dose-interruption, permanent discontinuation, or systemic immunosuppression due to immune-related AEs
9. Has primary central nervous system (CNS) tumors or brain or leptomeningeal metastasis.
10. Has human immunodeficiency virus (HIV) infection
11. Has active hepatitis B or C infection
12. Women who are pregnant or breastfeeding
13. Has an unwillingness or inability to comply with procedures required in this protocol
14. Is currently receiving any other anticancer or investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Part A: To determine the MTD or the RP2D of MPT-0118 | 1 cycle / 28 days
  The incidence and severity of treatment-emergent adverse events (TEAEs) qualifying as protocol-defined DLTs in Cycle 1 will guide the establishment of the protocol-defined RP2D and/or MTD.
Part B: To determine the MTD or the RP2D of MPT-0118 + pembrolizumab | 1 cycle / 28 days
  The incidence and severity of TEAEs qualifying as protocol-defined DLTs in Cycle 1 will guide the establishment of the protocol-defined RP2D and/or MTD.
Part C: Number of subjects with TEAEs as assessed by NCI-CTCAE v5.0 | Through study completion, an average of 1 year
  Incidence of TEAEs will be used to assess the safety of MPT-0118 + pembrolizumab
Part C: Objective response rate (ORR) based on RECIST v1.1 and iRECIST | Through study completion, an average of 1 year
Part C: Duration of response (DoR) based on RECIST v1.1 and iRECIST | Through study completion, an average of 1 year
Part C: Progression-free survival (PFS) based on RECIST v1.1 and iRECIST | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Part A and B: Maximum plasma concentration of MPT-0118 | 1 cycle / 28 days
Part A and B: ORR based on RECIST v 1.1 and iRECIST | Through study completion, an average of 1 year
Part A and B: DoR based on RECIST v 1.1 and iRECIST | Through study completion, an average of 1 year
Part A and B: PFS based on RECIST v 1.1 and iRECIST | Through study completion, an average of 1 year
Part C: Assessment of Overall Survival | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arthur DeCillis, MD, Study Director — Monopteros Therapeutics Inc.
Locations (5):
- United States (5):
  - St. John's Cancer Center, Santa Monica, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Di Pilato M, Gao Y, Sun Y, Fu A, Grass C, Seeholzer T, Feederle R, Mazo I, Kazer SW, Litchfield K, von Andrian UH, Mempel TR, Jenkins RW, Krappmann D, Keller P. Translational Studies Using the MALT1 Inhibitor (S)-Mepazine to Induce Treg Fragility and Potentiate Immune Checkpoint Therapy in Cancer. J Immunother Precis Oncol. 2023 Mar 3;6(2):61-73. doi: 10.36401/JIPO-22-18. eCollection 2023 May. PMID 37214210